CLINICAL TRIAL: NCT01113983
Title: A Clinical Trial of a Transcatheter Bioprosthetic Valve for Patients With Aortic Stenosis
Brief Title: PREVAIL-J - Transfemoral & Transapical Placement of Aortic Balloon Expandable Transcatheter Valves Trial (Japan)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EW-P-001
Record Dates: First submitted 2010-04-29; First posted 2010-04-30 (Estimated); Results first posted 2020-05-01 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Aortic Valve Stenosis
Keywords: SAPIEN XT Valve, Cardiovascular Disease, Valvular Heart Disease, Aortic Stenosis, Heart Valve Therapy, Transapical, Transcatheter, Transfemoral
MeSH Terms: conditions — Aortic Valve Stenosis; Cardiovascular Diseases; Heart Valve Diseases | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- TAVI - TF and TA approach (Experimental): Transcatheter aortic valve implantation and transfemoral/ transapical approach
  Interventions: Device: Transcatheter aortic valve implantation

INTERVENTIONS:
Device: Transcatheter aortic valve implantation — Transcatheter aortic valve implantation via transapical and transfemoral approach
  Other Names: SAPIEN XT; NovaFlex delivery system; Ascendra2 delivery system

SUMMARY:
A single arm, prospective multicenter non-randomized pivotal clinical trial evaluating the Edwards SAPIEN XT™ transcatheter heart valve (model 9300TFX), NovaFlex™ transfemoral delivery system, Ascendra2™ transapical delivery system and crimper accessories. The trial includes a premarket pivotal cohort to evaluate the system performance as well as a post market clinical follow-up phase involving long term follow-up of all patients to evaluate the safety of investigational devices up to 5 years.

DETAILED DESCRIPTION:
Purpose: To evaluate the safety and efficacy of THV-9300 for patients who have severe symptomatic aortic stenosis attributed to calcification and degeneration of a valve leaflet and for whom undergoing a surgery safely would be difficult.

Follow-up: Subject data collection will include clinical information at baseline and during the index procedure. Subjects will undergo clinical follow-up at discharge, 30 days, 6 months and annually for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were judged difficult to safely undergo AVR
* Severe senile degenerative aortic valve stenosis
* NYHA Functional Class II or greater
* Signed Informed Consent

Exclusion Criteria:

* Aortic valve is congenital unicuspid or bicuspid
* Annulus size between < 18 mm or > 25 mm
* LVEF < 20 %

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2010-04-01 (Actual); Primary Completion 2011-10 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yoshiki Sawa, MD, PhD, Principal Investigator — Osaka University Hospital
Locations (3):
- Japan (3):
  - Kurashiki Central Hospital, Kurashiki, Okayama-ken
  - Osaka University Hospital, Suita, Osaka
  - Sakakibara Heart Institute, Chōshi, Tokyo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sawa Y, Takayama M, Goto T, Takanashi S, Komiya T, Tobaru T, Maeda K, Kuratani T, Sakata Y; PREVAIL JAPAN Investigators. Five-Year Outcomes of the First Pivotal Clinical Trial of Balloon-Expandable Transcatheter Aortic Valve Replacement in Japan (PREVAIL JAPAN). Circ J. 2017 Jul 25;81(8):1102-1107. doi: 10.1253/circj.CJ-17-0111. Epub 2017 Mar 17. PMID 28321002
- [Derived] Watanabe Y, Hayashida K, Takayama M, Mitsudo K, Nanto S, Takanashi S, Komiya T, Kuratani T, Tobaru T, Goto T, Lefevre T, Sawa Y, Morice MC. First direct comparison of clinical outcomes between European and Asian cohorts in transcatheter aortic valve implantation: the Massy study group vs. the PREVAIL JAPAN trial. J Cardiol. 2015 Feb;65(2):112-6. doi: 10.1016/j.jjcc.2014.05.001. Epub 2014 Jun 11. PMID 24927855
- [Derived] Sawa Y, Takayama M, Mitsudo K, Nanto S, Takanashi S, Komiya T, Kuratani T, Tobaru T, Goto T. Clinical efficacy of transcatheter aortic valve replacement for severe aortic stenosis in high-risk patients: the PREVAIL JAPAN trial. Surg Today. 2015 Jan;45(1):34-43. doi: 10.1007/s00595-014-0855-y. Epub 2014 Mar 5. PMID 24595532

RESULTS

PARTICIPANT FLOW:
Groups:
- TAVI - TF Approach: Transcatheter aortic valve implantation and transfemoral approach
  Transcatheter aortic valve implantation: Transcatheter aortic valve implantation via transapical and transfemoral approach
- TAVI-TA Approach: Transcatheter aortic valve implantation - Transapical approach
Period: Overall Study
Arm/Group | TAVI - TF Approach | TAVI-TA Approach
Started | 37 | 27
Completed | 12 | 10
Not Completed | 25 | 17

BASELINE CHARACTERISTICS:
Groups:
- TAVI - TF Approach: Transcatheter aortic valve implantation and transfemoral approach
  Transcatheter aortic valve implantation: Transcatheter aortic valve implantation via transapical or transfemoral approach
- TAVI-TA Approach: Transcatheter aortic valve implantation - Transapical approach
  Transcatheter aortic valve implantation: Transcatheter aortic valve implantation via transapical or transfemoral approach
- Total: Total of all reporting groups
Arm/Group | TAVI - TF Approach | TAVI-TA Approach | Total
Number analyzed (Participants) | 37 | 27 | 64
Age, Continuous [Mean (Standard Deviation); unit: Years] | 83.2 (6.5) | 85.9 (5.3) | 84.3 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 18 | 42
  Male | 13 | 9 | 22
Height [Mean (Standard Deviation); unit: cm] | 151.10 (7.82) | 147.47 (8.55) | 149.57 (8.27)
NYHA III/IV [Number; unit: % of participants] — Measure Description: New York Heart Association (NYHA), functional classification of heart failure based on how much a patient is limited during physical activity. The rating ranges from I-IV, with the lowest as no limitations and the highest unable to carry on any physical activity without discomfort.
  % of participants | 40.5 | 48.1 | 43.8
NYHA II [Number; unit: % of Patients] — Measure Description: New York Heart Association (NYHA), functional classification of heart failure based on how much a patient is limited during physical activity. The rating ranges from I-IV, with the lowest as no limitations and the highest unable to carry on any physical activity without discomfort.
  % of Patients | 59.5 | 51.9 | 56.3
Arrhythmia [Number; unit: % of patricipants] | 56.8 | 37.0 | 48.4
Porcelain Aorta [Number; unit: % of Participants] | 13.5 | 22.2 | 17.2
Renal Disease [Number; unit: % of Participants] | 24.3 | 44.4 | 32.8

OUTCOME MEASURES:

1. Primary Outcome: Improvement of the AVA and NYHA Functional Classification
Description: Improvement of the aortic valve area (AVA) and New York Heart Association (NYHA) functional classification from baseline to 6 months after the procedure. NYHA functional classification of heart failure based on how much a patient is limited during physical activity. The rating ranges from I-IV, with the lowest (I) as no limitations and the highest (IV) unable to carry on any physical activity without discomfort. The AVA at 6 months > 1.0 cm2 indicates improvement. This outcome measure shows the percentage of patients that had an improvement in both NYHA Class and AVA.
Time Frame: 6 Months
Measure: Number; unit: % of participants
Arm/Group | TAVI - TF Approach | TAVI-TA Approach
Number analyzed (Participants) | 37 | 27
% of participants | 38.2 | 45.8

2. Secondary Outcome: Death
Description: Death Adverse Event Rate
Time Frame: 6 months
Measure: Number; unit: percentage of participants
Arm/Group | TAVI - TF Approach | TAVI-TA Approach
Number analyzed (Participants) | 37 | 27
percentage of participants | 5.4 | 18.5

ADVERSE EVENTS:
Time Frame: 6 Months
Arm/Group | TAVI - TF Approach | TAVI-TA Approach
All-Cause Mortality (participants affected / at risk) | 2/37 | 5/27
Serious Adverse Events (participants affected / at risk) | 25/37 | 27/27
Other Adverse Events (participants affected / at risk) | 19/37 | 13/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TAVI - TF Approach (N=37) | TAVI-TA Approach (N=27)
Acute adrenocortical insufficiency (Endocrine disorders) | 1 | 1
Anemia (Blood and lymphatic system disorders) | 0 | 1
Aortic Valve Replacement (Surgical and medical procedures) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Complete atrioventricular block (Cardiac disorders) | 2 | 6
Heart failure (Cardiac disorders) | 1 | 3
Cardiac tamponade (Cardiac disorders) | 1 | 0
Cardiopulmonary arrest (Cardiac disorders) | 2 | 0
Cerebral infarction (Vascular disorders) | 1 | 1
Suppurative cholangitis (Infections and infestations) | 0 | 1
Coronary occlusion (Cardiac disorders) | 0 | 1
Coronary stenosis (Cardiac disorders) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hepatic dysfunction (Hepatobiliary disorders) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Mastitis (Infections and infestations) | 0 | 1
Peripheral edema (General disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pneumonia (Infections and infestations) | 1 | 1
Sick sinus syndrome (Cardiac disorders) | 1 | 0
Hemorrhoid bleeding (Vascular disorders) | 2 | 3
Bleeding (Vascular disorders) | 2 | 3
Aortic rupture (Injury, poisoning and procedural complications) | 1 | 0
Obstructive airway disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tooth extraction (Surgical and medical procedures) | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1
Renal dysfunction (Renal and urinary disorders) | 1 | 0
Sepsis (Infections and infestations) | 0 | 1
Disuse syndrome (General disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Rotatory vertigo (Nervous system disorders) | 0 | 1
Study valve dislodge from aortic annulus (Surgical and medical procedures) | 1 | 0
Balloon contractile dysfunction (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TAVI - TF Approach (N=37) | TAVI-TA Approach (N=27)
Cystitis (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 0 | 1
Pseudomembranous colitis (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 1
Pseudomonas infection (Infections and infestations) | 0 | 1
Vocal cord polyp (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 1 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 8 | 11
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 0
Meniere's disease (Ear and labyrinth disorders) | 8 | 2
Aortic regurgitation (Cardiac disorders) | 1 | 8
Atrial fibrillation (Cardiac disorders) | 1 | 2
Atrioventricular block (Cardiac disorders) | 1 | 0
Complete atrioventricular block (Cardiac disorders) | 0 | 2
Left bundle branch block (Cardiac disorders) | 3 | 2
Right bundle branch block (Cardiac disorders) | 0 | 1
Heart failure (Cardiac disorders) | 1 | 2
Congestive heart failure (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1
Pulmonary congestion (Cardiac disorders) | 1 | 1
Tricuspid regurgitation (Cardiac disorders) | 0 | 1
Ventricular premature complex (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 1
Cerebellar infarction (Vascular disorders) | 0 | 1
Cerebral infarction (Vascular disorders) | 1 | 3
Intraoperative bleeding (Vascular disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Hepatic dysfunction (Hepatobiliary disorders) | 4 | 0
Contusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Diabetic nephropathy (Renal and urinary disorders) | 1 | 0
Renal dysfunction (Renal and urinary disorders) | 1 | 1
Peripheral edema (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Fever (General disorders) | 1 | 0
General health decline (General disorders) | 1 | 0
Elevation of CPK in blood (Investigations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No